CLINICAL TRIAL: NCT01507376
Title: Comparing the Efficacy of Urinary and Recombinant hCG on Oocyte Maturity for Ovulation Induction in Assisted Reproductive Techniques: a Randomized Clinical Trial
Brief Title: Comparing the Efficacy of Urinary and Recombinant Human Chorionic Gonadotropin (hCG) on Oocyte Maturity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Emb-012
Record Dates: First submitted 2011-09-14; First posted 2012-01-10 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2010-10

CONDITIONS: In Vitro Fertilization
Keywords: Ovulation induction; urinary; hCG; recombinant hCG
MeSH Terms: interventions — Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A: recombinant hCG(250 µg Ovitrell) (Experimental): 1- Group A consisted of 60 infertile women who received recombinant hCG(250 µg Ovitrelle)
  Interventions: Drug: recombinant hCG
- B: recombinant hCG(500 µg Ovitrell) (Experimental): 2- Group B consisted of 60 infertile women who received recombinant hCG(500 µg Ovitrelle)
  Interventions: Drug: recombinant hCG
- C: urinary hCG (Experimental): 3- Group C consisted of 60 infertile patients received 10,000 IU urinary hCG
  Interventions: Drug: urinary hCG

INTERVENTIONS:
Drug: recombinant hCG — recombinant hCG(250 µg Ovitrell)
  Arms: A: recombinant hCG(250 µg Ovitrell)
Drug: recombinant hCG — recombinant hCG(500 µg Ovitrell)
  Arms: B: recombinant hCG(500 µg Ovitrell)
Drug: urinary hCG — 10,000 IU urinary hCG
  Arms: C: urinary hCG

SUMMARY:
This study is a prospective randomized clinical trial to compare the efficacy of the urinary and recombinant hCG on oocyte quality for ovulation induction in women undergoing IVF/ICSI.

DETAILED DESCRIPTION:
The study population comprised of all infertile patients aged 20-37 years which underwent of in-vitro fertilization in royan institute, Tehran Iran.

In this study all patients were treated with a long stimulation protocol in which GnRH-analogue (Buserelin subcutaneous, 0.5cc daily) was given as a pre-treatment and recombinant FSH (rFSH) administration was started when pituitary desensitization was confirmed. From the 7th day of stimulation in both groups, daily monitoring of follicle size by ultrasound was performed and the dose of rFSH was adjusted according to the response of each patient. When at least two follicles > 18 mm diameter were seen, ovulation was triggered with hCG and patients allocated into three different study groups as per the following:

1. Group A consisted of 60 women who received recombinant hCG(250 µg Ovitrelle)
2. Group B consisted of 60 women who received recombinant hCG(500 µg Ovitrelle)
3. Group C consisted of 60 patients received 10,000 IU urinary hCG Oocyte retrieval performed about 34-36 hours after hCG administration and then oocytes were assessed for nuclear maturity. Embryos transferred 2-3 days thereafter.

Data collection will be performed by using questionnaire to be filled as per the available records and laboratory results. Data analysis will be done through descriptive and perceptive statistical methods by using SPSS software version 16 for windows.

ELIGIBILITY:
Inclusion Criteria:

* Indication for IVF/ICSI and Long Protocol ovarian stimulation
* Age 20-37
* Body mass index (BMI) ≤ 30 kg/m2
* Regular menstrual cycles of 25-35 days
* Tubal or male factor
* Existence of both ovary and normal uterine cavity
* Basal FSH≥10
* Physical health

Exclusion Criteria:

* Poly Cystic Ovarian Syndrome patients
* Contraindications of gonadotropins administration
* Poor response to ovulation induction in recent cycle

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of mature oocytes | Up to1 hour after oocyte retrieval
  evaluation the effect of recombinant hcg on number of oocytes up to 1 hour after oocytes retrieval

SECONDARY OUTCOMES:
number of retrieved oocytes per number of aspirated follicles proportion | up to 1 hour after oocyte retrieval
  Evaluation the effect of recombinant hCG to retrieve oocytes per number of aspirated follicles proportion
fertilization rate | in 1 day after oocyte retrieval
  Evaluation the effect of recombinant hCG on fertilization rate in 1 day after oocyte retrieval
implantation rate | 4 weeks after embryo transfer
  Evaluation the effect of recombinant hCG on implantation rate 4 weeks after embryo transfer
OHSS occurrence rate will be compared between three groups | from embryo transfer day up to pregnancy test
  Evaluation the effect of recombinant hCG on OHSS occurrence rate will be compared between three groups
chemical pregnancy rates | 2 weeks after embryo transfer
  Evaluation the effect of recombinant hCG on chemical pregnancy rates 2 weeks after embryo transfer
clinical pregnancy rates | 4 weeks after embryo transfer
  Evaluation the effect of recombinant hCG on clinical pregnancy rates 4 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Taraneh Madani, MD, Study Director — gynecology scientist; Ladan Mohmmadi yeganeh, MSc, Principal Investigator — Investigator
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Madani T, Mohammadi Yeganeh L, Ezabadi Z, Hasani F, Chehrazi M. Comparing the efficacy of urinary and recombinant hCG on oocyte/follicle ratio to trigger ovulation in women undergoing intracytoplasmic sperm injection cycles: a randomized controlled trial. J Assist Reprod Genet. 2013 Feb;30(2):239-45. doi: 10.1007/s10815-012-9919-3. Epub 2012 Dec 29. PMID 23274511
- See also: Related Info — http://www.royaninstitute.org/cmsen/index.php